CLINICAL TRIAL: NCT02874066
Title: Paritaprevir/Ritonavir/Ombitasvir Plus Dasabuvir for Treatment-Naive and Treatment-Experienced Non-Cirrhotic Patients With Hepatitis C Virus Genotype 1b Receiving Hemodialysis
Brief Title: PrOD for Non-Cirrhotic Patients With HCV-1b Receiving Hemodialysis
Acronym: PIVOTAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201606016MIPC
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis Viruses
Keywords: Hepatitis C virus; Hemodialysis; Direct acting antiviral agents
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTV/r/OBV/DSV (Experimental): Paritaprevir/ritonavir/ombitasvir (PTV/r/OBV, 75mg/50mg/12.5mg per tablet, Viekirax): 2 tablets per os per day Dasabuvir (DSV, 250 mg per tablet, Exviera): 1 tablet per os twice per day Treatment duration: 12 weeks
  Interventions: Drug: PTV/r/OBV/DSV

INTERVENTIONS:
Drug: PTV/r/OBV/DSV — Viekirax/Exviera for 12 weeks
  Other Names: Viekirax/Exviera

SUMMARY:
Hepatitis C virus (HCV) infection is common in patients receiving hemodialysis. The uptake of antiviral therapy for these patients is limited in the era of interferon (IFN) plus ribavirin (RBV), probably because the sustained virologic response (SVR) rates are low and the risk of treatment-related adverse events (AEs) are high. In the era of IFN-free direct acting antiviral agents (DAAs), several studies have indicated high rates of SVR and excellent safety profiles to treat patients with severe renal impairment. With regard to ombitasvir/paritaprevir/ritonavir plus dasabuvir (PrOD) treatment, a phase 2 study (RUBY-1) study has shown 90% of SVR in treatment-naive HCV-1 patients with chronic kidney disease (CKD) stage 4 or 5. Among the HCV-1b patients, who received PrOD for 12 weeks, all 7 patients achieved SVR. Although the data confirmed the excellent safety and efficacy in HCV-1b patients with severe renal impairment, the patient number was small and the data with regard to treatment-experienced patients was lacking. Therefore, we aimed to evaluated the safety and efficacy of ProD for 12 weeks in treatment-naive and treatment-experienced HCV-1b patients receiving hemodialysis.

DETAILED DESCRIPTION:
Overview Hepatitis C virus (HCV) infection remains a major co-morbidity in hemodialysis patients. The incidence and prevalence rates of HCV infection in hemodialysis patients are much higher than those in the general population, and are attributed to high rates of nosocomial HCV transmission. With regard to HCV genotype distribution, HCV genotype 1 (GT-1) infection is the most prevalent type of infection worldwide and the genotype distribution in HCV-infected individuals receiving hemodialysis (HD) is similar to that observed in HCV-infected individuals with normal renal function.Compared to non-HCV infected hemodialysis patients, HCV-infected patients have increased risks of liver-related morbidity and mortality.10 Although HCV-infected hemodialysis patients who receive renal transplantation have survival advantages over those who remain on maintenance dialysis, these patients still have poor patient and graft survival, as well as have poor responses to interferon (IFN)-based therapy. In contrast, hemodialysis patients who eradicate HCV infection have improved biochemical, virologic and histologic responses, whether on maintenance dialysis or after renal transplantation.

Clinical experience of IFN-based Therapy Approximately one third of hemodialysis patients with chronic HCV infection achieve sustained virological response (SVR) by conventional IFN or peginterferon monotherapy. In addition 18-30% of patients receiving IFN-based monotherapy prematurely discontinued treatment due to adverse events (AEs). Although the addition of ribavirin to IFN further improves the SVR rate in HCV-infected patients with normal renal function, ribavirin has been considered contraindicated to treat HCV-infected hemodialysis patients because of concern for life-threatening hemolytic anemia. Recently, pilot studies have indicated the feasibility of adding low-dose ribavirin (200 mg three times per week to daily 400 mg, adjusted to achieve a target concentration of 10-15 μmol/L), to IFN for treatment of HCV-infected hemodialysis patients. Generally, the SVR rate and the premature discontinuation rate due to null-response, severe anemia, and/or heart failure for combination therapy are 56% and 22%, respectively.Based on these small-scale studies, low-dose ribavirin (daily 200 mg) was approved in August 2011 by the U.S. Food and Drug Administration to treat HCV-infected hemodialysis patients.Two recent well-conducted randomized control studies to compare the efficacy and safety of combination therapy with peginterferon alfa-2a (135 μg/week) plus low-dose ribavirin (RBV) (200 mg/day) or monotherapy with peginterferon (135 μg/week) for 48 and 24 weeks in treatment-naïve HCV GT-1 and GT-2 infected individuals receiving hemodialysis showed that the SVR rates of combination therapy groups were greater than those of monotherapy groups (64% versus 34%, p < 0.001 for HCV GT-1; 74% versus 44%, p < 0.001 for HCV GT-2), respectively. Although the SVR rate of combination therapy with peginterferon plus low-dose ribavirin is higher than that of peginterferon monotherapy. About 70-75% of these patients experienced clinically significant anemia which needed high dose of erythropoiesis stimulating agents (ESAs) to keep the hemoglobin level within the safety range. Although telaprevir (TVR)-based triple therapy has been used to treat 4 HCV-1 patients receiving hemodialysis who were not responsive to prior peginterferon plus RBV with good efficacy, the added on-treatment adverse events (AEs) and the pill burden precluded the widespread use of this agent.

Clinical experience of IFN-free therapy by ombitasvir/paritaprevir/ritonavir plus dasabuvir in HCV GT-1 patients The recent introduction of IFN-free direct acting antiviral agents (DAAs) has made a paradigm shift with regard to the medical treatment for HCV-infected individuals, based on the excellent efficacy and safety in ordinary patients. Among the various IFN-free DAA regimens, treatment with ombitasvir/paritaprevir/ritonavir plus dasabuvir (PrOD) has been approved in 2014 to treat patients with chronic HCV GT-1 infection. Treatment with PrOD plus weight-based ribavirin for 12 weeks achieved an SVR12 rate of 96.2% and 96.3% in treatment-naïve and treatment-experienced non-cirrhotic HCV GT-1 patients, respectively (SAPPHIRE-I and SAPPHIRE-II). Furthermore, the SVR12 rates in those with GT-1a and GT-1b were 95.3% and 98.0% in treatment-naïve patents, and 96.0% and 96.7% in treatment-experienced patients, respectively. Among treatment-experienced HCV-1 patients, the SVR rates of PrOD plus RBV were comparable in those with various prior treatment responses by peginterferon plus RBV (relapse: 95.3%; partial response: 100%, null response: 95.2%).36 Among treatment-naïve and treatment-experienced compensated cirrhotic HCV GT-1 patients, treatment with PrOD plus RBV for 12 or 24 weeks achieved and SVR rate of 91.8% and 95.%, respectively (TURQUOISE-II).37 The SVR12 rates in HCV GT-1b cirrhotic patients were similar in those receiving 12 and 24 weeks of treatment (98.5% versus 100%); the SVR12 rate in HCV GT-1a cirrhotic patients receiving 24 week of treatment was greater than those receiving 12 weeks of treatment (94.2% versus 88.6%), particularly for prior non-responders to peginterferon plus RBV (92.9% versus 80%). The PEARL-III and PEARL-IV studies compared the SVR12 rates in treatment-naïve non-cirrhotic HCV GT-1b and HCV GT-1a patients receiving PrOD with/without RBV for 12 weeks.37 The SVR12 rate of PrOD without RBV was similar to that of PrOD with RBV in HCV GT-1b patients (99.0% versus 99.5%). However, the SVR12 rate in HCV GT-1a patients receiving PrOD with RBV was marginally higher than those receiving PrOD without RBV (97.0% versus 90.2%). The PEARL-II study further confirmed that in treatment-experienced non-cirrhotic HCV GT-1b patients, treatment with PrOD without RBV for 12 weeks had comparable SVR12 rate to PrOD with RBV therapy (100% versus 96.6%). In TURQUOISE-III study, PrOD without RBV for 12 weeks achieved an SVR12 rate of 100% in treatment-naïve and treatment-experienced compensated cirrhotic HCV GT-1b patients. With regard to safety, PrOD with/without RBV showed excellent safety profiles with few patients experiencing serious adverse events (SAEs) and prematurely treatment discontinuation. The constitutional AEs in patients receiving PrOD based treatment showed were slightly higher than those receiving placebo. Furthermore, most of these symptoms were mild in grades. About 5% of the non-cirrhotic patients and about 8% of the cirrhotic patients receiving PrOD plus RBV had an on-treatment hemoglobin level of < 10 g/dL; and none of the non-cirrhotic patients and about 2% of the compensated cirrhotic patients receiving PrOD had an on-treatment hemoglobin level of < 10 g/dL, respectively.35-40 In addition, the on-treatment AST/ALT elevation of more than 5 times the upper limit of normal (ULN) were 0.6%-1.7% and 0.5% in non-cirrhotic patients receiving PrOD with and without RBV; and were 2.9% and 2.0% in compensated cirrhotic patients receiving PrOD with and without RBV, respectively. The on-treatment total bilirubin elevation of more than 3 times ULN were 2.4%-5.7% and 0.5% in non-cirrhotic patients receiving PrOD with and without RBV; 13.5% and 0% in compensated cirrhotic patients receiving PrOD with and without RBV, respectively.35-40 Based on the above evidence, treatment with PrOD for 12 weeks is recommended for treatment-naïve and treatment-experienced HCV GT-1b patients, regardless of cirrhosis or not. Treatment with PrOD plus RBV for 12 weeks is recommended for HCV GT-1a patients, except for compensated cirrhotic HCV GT-1a null responders to prior therapy where treatment with PrOD plus RBV for 24 weeks is recommended.

Clinical experience of IFN-free therapy by ombitasvir/paritaprevir/ritonavir plus dasabuvir in HCV GT-1 patients with severe renal impairment or end-stage renal disease (ESRD) The pharmacokinetic (PK) study of ombitasvir, paritaprevir, ritonavir, and dasabuvir was evaluated in 24 subjects with normal renal function, and with mild, moderate or severe renal impairment (each arm 6 patients). Compared to subjects with normal renal function, the area under the curves (AUCs) in subjects with mild renal impairment were comparable for ombitasvir, 20% higher for paritaprevir and dasabuvir, and 42% higher for ritonavir; the AUCs in subjects with moderate renal impairment were comparable for ombitasvir, 37% higher for paritaprevir and dasabuvir, and 80% higher for ritonavir; the AUCs in subjects with severe renal impairment were comparable for ombitasvir, 50% higher for paritaprevir and dasabuvir, and 114% higher for ritonavir. All patients were well tolerated for PrOD treatment except for mild AEs, including nausea, myalgia, and catheter-site erythema, encountered in 1 subject with moderate renal impairment. Based on the PK study, the changes of the drug exposure were not clinically relevant and the doses of PrOD do not require adjustment.

The phase 3b RUBY-I study evaluated the safety and efficacy of PrOD with RBV and PrOD without RBV for 12 weeks in 13 and 7 HCV GT-1a and HCV GT-1b treatment-naïve non-cirrhotic patients with severe renal impairment or ESRD. The interim safety analysis showed that no patients had study drug discontinuation, no treatment-related serious adverse events (SAEs) and no clinically significant changes in markers of liver or kidney function. With regard to efficacy, 14 of the 20 patients completed 12 weeks of treatment and all of them achieved end-of-treatment virologic response (EOTVR). Ten patients (8 in GT-1a and 2 in GT-1b) completed post-treatment follow-up for 4 weeks and all achieved SVR4. Furthermore, 2 HCV GT-1a patients completed post-treatment follow-up for 12 weeks and all achieved SVR12.

Rationale of the study design Although peginterferon monotherapy and combination therapy with peginterferon plus low-dose RBV for 24-48 weeks have been evaluated in many studies, the efficacy for the treatment regimens were only modest (SVR rate about 60%). In addition, the on-treatment AEs and SAEs by IFN-based therapies were frequently encountered in HCV-infected patients receiving hemodialysis. Of note was the pronounced on-treatment hemoglobin level decrease in patients receiving combination therapy by peginterferon plus low-dose RBV, necessitating significant RBV dose reduction and high-dose erythrocyte stimulating agent (ESA) support.

By receiving IFN-free DAA therapies, HCV-infected patients have excellent SVR rates, low on-treatment SAE and AE rates, shorter treatment duration, and low pill burdens. The PK study of ombitasvir, paritaprevir, ritonavir and dasabuvir proves the excellent safety profiles and dose adjustment are not needed for PrOD regimen in subjects with various degrees of renal impairment. The interim analysis of RUBY-I study showed the excellent on-treatment and off-therapy antiviral effects in HCV GT-1a and GT-1b infected patients receiving PrOD plus low-dose RBV and PrOD, respectively. However, all the patients enrolled in the RUBY-I study were treatment-naïve and were non-cirrhotic. Furthermore, only 7 patients in the RUBY-I study were HCV GT-1b patients. Based on the excellent safety and efficacy profiles of PrOD treatment for HCV GT-1b infected patients with normal renal function, we aim to evaluate the safety and efficacy of PrOD for 12 weeks in treatment-naïve and treatment-experienced HCV GT-1b non-cirrhotic patients receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 20 to 70 yeas
* Male or female
* Body mass index (BMI) 18.5-35.0 kg/m2
* Chronic HCV infection, defined as patients who meet as least one of the two following criteria

  1. Anti-HCV antibody (Abbott HCV enzyme-linked immunosorbent assay [EIA] 2.0, Abbott Laboratories, Abbott Park, Illinois, USA) or HCV RNA > 1,000 IU/mL for at least 6 months before screening
  2. Positive HCV RNA > 1,0000 IU/mL (Cobas TaqMan HCV Test v2.0, Roche Diagnostics Gesellschaft mit beschränkter Haftung [GmbH], Mannheim, Germany, low limit of quantification (LLOQ): 25 IU/mL) at the time of screening with a liver biopsy consistent with chronic HCV infection
* HCV GT-1b infection (Abbott RealTime HCV genotyping II, Abbott Molecular Inc. Illinois, USA)
* Treatment-naïve or treatment-experienced (including patients who relapsed, who had virological breakthrough, or who were null-responsive to IFN-based therapies)
* HCV RNA > 10,000 IU/mL at screening
* Absence of cirrhosis with documented results of one of the following criteria:

  1. Liver biopsy within 24 months prior to or during screening demonstration the absence of cirrhosis, e.g. METAVIR score ≤ 3 or Ishak score ≤ 4.
  2. A screening transient elastography (Fibroscan) result of < 12.5 kilopascal (kPa)
  3. A screening Fibrosis Index Based on 4 markers (FIB-4) of ≤ 1.45 and Aspartate Aminotransferase to Platelet Ratio Index (APRI) of ≤ 2
  4. Subjects with non-qualifying FIB-4/APRI or Fibroscan result may only be enrolled if they have a qualifying liver biopsy within 24 months prior to or during screening
* Estimated glomerular filtration (eGFR) rate < 15 mL/min/1.73m2 as assessed by modified of diet in renal disease (MDRD) equation, and receiving regular hemodialysis

Exclusion Criteria:

* HCV infection other than HCV GT-1b
* Hepatitis B virus (HBV) or HIV co-infection
* Presence of cirrhosis (Child-Puge class A, B or C)
* Any primary cause of liver disease other than chronic HCV infection, including but not limited to the following

  1. Hemochromatosis
  2. Alfa-1 antitrypsin deficiency
  3. Wilson's disease
  4. Autoimmune hepatitis
  5. Alcoholic liver disease
  6. Drug-induced hepatitis
* Screening laboratory analyses showing any of the following results

  1. Hemoglobin (Hb) level < 10 g/dL
  2. Absolute neutrophil count (ANC) < 1,500 cells/μL
  3. Platelet count < 60,000 cells/mm3
  4. International normalized ratio (INR) > 2.0
  5. Albumin (Alb) < 2.8 g/dL
  6. Bilirubin (Bil) > 3.0 mg/dL
  7. Alanine aminotransferase (ALT) > 5X upper limit of normal (ULN)
  8. Aspartate aminotransferase (AST) > 5X upper limit of normal (ULN)
  9. Serum alfa-fetoprotein (AFP) > 100 ng/mL
* Presence of hepatocellular carcinoma (HCC) on imaging studies such as computed tomography (CT) scan or magnetic resonance imaging (MRI)
* History of malignancy (except cutaneous melanoma) within 5 years at the screening
* Organ transplantation other than cornea and hair (prior renal transplantation with graft failure not included)
* Prior exposure to investigational agents for HCV (direct acting antiviral agents, host-targeting agents, or therapeutic vaccines)
* Pregnancy
* Unwilling to have contraception during the study period [12] Unwilling to provide informed consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, PhD, Study Director — National Taiwan University Hospital
Locations (8):
- Taiwan (8):
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital, Chiayi City
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei City Hospital, Ren-Ai Branch, Taipei
  - Tri-Service General Hospital, National Defense Medical Center, Taipei

IPD SHARING:
Plan to Share IPD: No
Confidential of the individual participant data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 64 patients screened, 18 patients excluded
Period: Overall Study
Arm/Group | PTV/r/OBV/DSV
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PTV/r/OBV/DSV
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 58 [37 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Taiwan | 46
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 46
HCV RNA [Median (Full Range); unit: Log10 IU/mL] — Log10 IU/mL
  Log10 IU/mL | 5.60 [2.96 to 7.22]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virologic Response (SVR12)
Description: Number of participants with undetectable serum HCV RNA 12 weeks off therapy (treatment period 12 weeks)
Time Frame: 24 weeks
Population: Patients who received at least one dose of PTV/r/OBV/DSV
Measure: Count of Participants; unit: Participants
Arm/Group | PTV/r/OBV/DSV
Number analyzed (Participants) | 46
Participants | 46

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Event (AE)-Related Withdrawal Rate
Description: Number of participants with treatment-emergent adverse event (AE)-related withdrawal rate during the study
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PTV/r/OBV/DSV
Number analyzed (Participants) | 46
Participants | 0

3. Secondary Outcome: Number of Participants With Sustained Virologic Response (SVR24)
Description: Number of participants with undetectable serum HCV RNA 24 weeks off therapy (treatment period 12 weeks)
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PTV/r/OBV/DSV
Number analyzed (Participants) | 46
Participants | 46

4. Secondary Outcome: Number of Participants With Rapid Virologic Response (RVR)
Description: Number of participants with undetectable serum HCV RNA at week 4 of treatment
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PTV/r/OBV/DSV
Number analyzed (Participants) | 46
Participants | 46

5. Secondary Outcome: Number of Participants With End-of-treatment Virological Response (EOTVR)
Description: Number of participants with undetectable serum HCV RNA at week 12 of treatment
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PTV/r/OBV/DSV
Number analyzed (Participants) | 46
Participants | 46

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | PTV/r/OBV/DSV
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 2/46
Other Adverse Events (participants affected / at risk) | 19/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTV/r/OBV/DSV (N=46)
Acute gastroenteritis (Gastrointestinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTV/r/OBV/DSV (N=46)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9)
Fatigue (General disorders) | 7 (7)
Upper respiratory tract infectioin (Infections and infestations) | 3 (3)

LIMITATIONS AND CAVEATS:
This study did not evaluate Child-Pugh A cirrhotic HCV-1b patients receiving hemodialysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT02874066/Prot_SAP_000.pdf